CLINICAL TRIAL: NCT05838209
Title: Effect of Ozone Oil After Non-surgical Periodontal Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Gabriela Alessandra da Cruz Galhardo Camargo, Clinical Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE 89966418.8.0000.5626
Record Dates: First submitted 2023-04-05; First posted 2023-05-01 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Periodontal Diseases
Keywords: Periodontitis, Periodontal treatment, diabetes
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This is a prospective clinical randomized controlled, split mouth designed, doble blinded study.
Who Masked: Participant, Care Provider
Masking Description: Participants - The randomization performed will use the coin heads or tails method, Investigators -Two treatments at randomly chosen sites separate in two groups: Ozone oil use as an adjunctive of scaling and root planing and saline solution 0.09%, as a control, associate as an adjunctive of scaling and root planing. Ultrasonic scaler and Gracey curets use to remove all calculus and biofilms during scaling and root planing. The oils are numbere syringes labeled 1 and 2 for blinded applications, and 1 ml of each oil were administrated in a previous selected site. After removing baseline samples of biofilm, the scaling and root planing were performed using ultrasonic devices and manual Gracey curettes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Scaling and root planing + saline solution gel (control) will be adminster at probing depth > 5mm.
  Interventions: Drug: Control
- Test (Active Comparator): Scaling and root planing + Ozone Oil will be adminster at probing depth > 5mm.
  Interventions: Drug: test

INTERVENTIONS:
Drug: test — Ozone oil used as an adjunctive of scaling and root planing and control,
  Arms: Test
Drug: Control — saline solution 0.09% used as an adjunctive as scaling and root planing
  Other Names: Placebo Control
  Arms: Control

SUMMARY:
The goal of this clinical trial is to evaluate the use of ozone oil as an adjunctive of non-surgical periodontal treatment (NSPT) on diabetics type 2 patients (DM2) compared to control group with chronic periodontal disease.

The principal question is to evaluate if the ozone oil could improve periodontal clinical parameters.

Thirty-two sites of 16 diabetics type 2 patients (DM2) with moderate to advanced periodontal disease containing two sites with periodontal pocket depth (PPD) of > 5 mm were selected.

The treatment was distributed in 2 groups in the split mouth design: Control- scaling and root planing + saline solution (control) and Test - scaling and root planning + ozone oil

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis
* Systemic type 2 diabetes

Exclusion Criteria:

* Hypersensitivity to ozone oil
* Osteoporosis types I and II
* Alcoholism
* Immunosuppressio
* Pregnant and lactating
* Physical/emotional stress drugs
* Use of antibiotics, anti-inflammatories and hormone
* Oral candidiasis
* Received periodontal treatment in the last six months prior to the procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — patients over 18 years old
Enrollment: 16 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Plaque Index | baseline
  Percentage
Gingival Index | baseline
  Percentage
Probing Depth | baseline
  mm
clinical attachment level | baseline
  mm

SECONDARY OUTCOMES:
Plaque Index | 3 months
  Percentage
Gingival Index | 3 months
  Percentage
Probing Depth | 3 months
  mm
clinical attachment levels | 3 months
  mm

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriela Alessandra da Cruz Galhardo Camargo, Nova Friburgo, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mauri-Obradors E, Merlos A, Estrugo-Devesa A, Jane-Salas E, Lopez-Lopez J, Vinas M. Benefits of non-surgical periodontal treatment in patients with type 2 diabetes mellitus and chronic periodontitis: A randomized controlled trial. J Clin Periodontol. 2018 Mar;45(3):345-353. doi: 10.1111/jcpe.12858. Epub 2018 Jan 19. PMID 29265454